CLINICAL TRIAL: NCT05162911
Title: Implementing Tobacco Use Treatment in HIV Clinics in Vietnam
Brief Title: Implementing Tobacco Use Treatment in HIV Clinics Vietnam
Acronym: Vquit
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: i19-01783
Record Dates: First submitted 2021-11-10; First posted 2021-12-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-05

CONDITIONS: Tobacco Use
Keywords: Tobacco Use; Implementation Science
MeSH Terms: conditions — Tobacco Use | interventions — corticosteroid hormone-induced factor; Insemination, Artificial, Heterologous; Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ask, Advise, Assist (AAA) and Refer. (Active Comparator): Patients will receive Ask, Advise, Assist (AAA) and refer to the quitline as the intervention.
  Interventions: Behavioral: Ask, advise, Assist and refer to the Quitline
- AAA plus referral to onsite counselor (Counsel). (Active Comparator): Patients will receive Ask, Advise, Assist plus referral to onsite counselor.
  Interventions: Behavioral: Ask, advise, Assist and referral to onsite counselor
- AAA+Counsel+N (Nicotine gum). (Active Comparator): Patients will receive Ask, Advise, Assist, plus referral to onsite counselor and nicotine gum.
  Interventions: Behavioral: Ask, advise, Assist and referral to onsite counselor and NRT

INTERVENTIONS:
Behavioral: Ask, advise, Assist and refer to the Quitline — A nurse will ask, advise, assist and refer patient to the Quitline
  Arms: Ask, Advise, Assist (AAA) and Refer.
Behavioral: Ask, advise, Assist and referral to onsite counselor — A nurse will ask, advise, assist and refer patient to a counselor
  Arms: AAA plus referral to onsite counselor (Counsel).
Behavioral: Ask, advise, Assist and referral to onsite counselor and NRT — A nurse will ask, advise, assist and refer patient to a counselor and provide nicotine replacement therapy in the form of gum
  Arms: AAA+Counsel+N (Nicotine gum).

SUMMARY:
The primary objective of this study is to conduct a 3-arm randomized controlled trial (RCT) that compares the effectiveness of three multi-component interventions that are embedded in HIV outpatient clinics (OPCs): 1)3As+Referral to the national quitline: Ask about tobacco use, Advise to quit, Assist with brief counseling and Refer to Viet Nam's national Quitline; 2) AAA+ +Counsel (Counsel=6-session cessation counseling intervention adapted for patients living with HIV/AIDS (PLWH) and delivered by a trained, onsite nurse; and 3) AAA+Counsel+N (N=nicotine replacement therapy (NRT)). The main outcome is biochemically validated 6-months smoking abstinence. The investigators will recruit and randomize 672 patients across 13 outpatient clinics (OPCs) (48 per site, 16 per arm). The investigators will also recruit 75-nonsmokers to participate in a single survey to assess food safety. Therefore, the total sample = 747 patients.

DETAILED DESCRIPTION:
This research has three phases. For Aim 1 the investigators will conduct a formative assessment to inform further modifications to the intervention components. Participants in Aim 1 will be patients of the outpatient clinics (OPC) or health care providers who work there. Patients who use tobacco will be asked to participate in individual interviews (n=24 ). The investigators will conduct key informant interviews with health care providers from 3 OPCs (n=28) to adapt the intervention to the OPC clinical context. The investigators will then conduct a pilot test of ARM 1 and 3 in one OPC with 16 patients. The recruitment and enrollment process will be the same as described for Aim 2. For Aim 2 the investigators will conduct a three-arm randomized controlled trial (RCT) to compare the effectiveness of three interventions aimed at increasing tobacco cessation rates among people living with HIV/AIDS (PLWH). Patients (n=672) will be recruited and enrolled from the 13 OPCs. All enrolled patients will complete a baseline survey in person. This survey will be administered once eligibility is established and consent is obtained. The consent and survey will last 30 minutes. Follow up surveys will occur at 3-, -6 and 12-months after enrollment. Follow up surveys will be conducted by telephone. At 6-months follow up, patients who report smoking abstinence will be asked to come in person to the OPC and will complete a carbon monoxide test to validate self-report. The investigators will conduct baseline, 12 and 18 month surveys with all health care providers in the study sites in person (n=98). For Aim 3 the investigators will conduct a post intervention (12-month) assessment of factors associated with implementation effectiveness and potential for sustainability. This includes repeating the health care provider surveys and Key informant interviews. The investigators will conduct baseline, 12 and 18 month surveys with all health care providers in the study sites in person (n=98). For Aim 4 the investigators will enroll 75 more patients who are non-smokers for a total of (n=747) patients and assess the relationship between food insecurity and tobacco use among PLWH (75 smokers and 75 non-smokers), which includes administering the Household Food Insecurity Access Scale (HFIAS) survey to patients at baseline and 6-months.

ELIGIBILITY:
Inclusion Criteria:

* patients in the HIV OPCs
* current tobacco users
* patients who live in Hanoi
* patients reachable by phone

Exclusion Criteria:

* patients for whom there is a need for precaution in using NRT will be excluded
* patients with recent myocardial infarction (2 weeks)
* patients serious underlying arrhythmias
* patients who are pregnant or nursing
* patients are unable to demonstrate capacity for consent
* patients already enrolled in a tobacco use treatment program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Carbon test at 6-months of smoking abstinence | 6-months smoking abstinence
  biochemically validated 6-months smoking abstinence will be measured using expired-air carbon monoxide reading equal to or less than 8 ppm (CO < 8 ppm). The scale is 0-50ppm, where the lowest values represent less CO levels, which indicate a patient is not smoking, and the highest values represent higher CO levels indicating a patient is actively smoking.

SECONDARY OUTCOMES:
Factors that may influence tobacco cessation, and sustainability of the interventions tested | 18 months
  Using questionnaires measure health care setting, provider, and patient level factors that may influence tobacco cessation, and sustainability of the interventions tested.

CONTACTS AND LOCATIONS:
Locations (1):
- Nam Nguyen, Hanoi, Nam Tu Liem, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shelley D, Alvarez GG, Nguyen T, Nguyen N, Goldsamt L, Cleland C, Tozan Y, Shuter J, Armstrong-Hough M. Adapting a tobacco cessation treatment intervention and implementation strategies to enhance implementation effectiveness and clinical outcomes in the context of HIV care in Vietnam: a case study. Implement Sci Commun. 2022 Oct 17;3(1):112. doi: 10.1186/s43058-022-00361-8. PMID 36253834

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT05162911/Prot_SAP_000.pdf